CLINICAL TRIAL: NCT01152073
Title: A Multicenter Study Of Nutraceutical Drinks For Cholesterol (Evaluating Effectiveness and Tolerability)
Brief Title: A Study Of Nutraceutical Drinks For Cholesterol (Evaluating Effectiveness and Tolerability)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Healthy Drink Discoveries, Inc. (Other)
Responsible Party: Principal Investigator, Dr. Mitchell Karl, Principal Investigator, Healthy Drink Discoveries, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 2009.35
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Hyperlipidemia
Keywords: Cholesterol; Statin; Nutraceuticals; Niacin; Hyperlipidemia; Liquid
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Study participants whose drink formulation contains no active ingredients but will appear and taste similar to the two other formulations. This will form the control formulation
  Interventions: Dietary Supplement: Placebo
- Second Formulation (Active Comparator): Study participants' drink formulation will include Red Yeast Rice 600mg, Niacin 12.5mg, Phytosterol esters 650mg, L-Carnitine 150mg, vitamin C 500mg, and Co-Q-10 25mg.
  Interventions: Dietary Supplement: Second Formulation
- Third Formulation (Active Comparator): The third formulation will be identical to the second, but without the Red Yeast Rice.
  Interventions: Dietary Supplement: Third Formulation

INTERVENTIONS:
Dietary Supplement: Placebo — Each subject will be expected to consume a twice daily drink of approximately 4 ounces per serving taken with the morning and evening meals for a total of 8 weeks. Each bottle will contain two servings.
  Arms: Placebo
Dietary Supplement: Second Formulation — Each subject will be expected to consume a twice daily drink of approximately 4 ounces per serving taken with the morning and evening meals for a total of 8 weeks. Each bottle will contain two servings.
  Arms: Second Formulation
Dietary Supplement: Third Formulation — Each subject will be expected to consume a twice daily drink of approximately 4 ounces per serving taken with the morning and evening meals for a total of 8 weeks. Each bottle will contain two servings.
  Arms: Third Formulation

SUMMARY:
Great controversy exists about the feasibility and safety of a product that can be employed for self-directed cholesterol reduction. The position that self-directed cholesterol lowering could lead those that do not need lower cholesterol to take the product is likely unfounded. This is because there is no convincing evidence to suggest that there are cholesterol levels so low that a lower one would not be beneficial or conversely be dangerous. Ample evidence exists that cholesterol causes cardiovascular disease and that lower cholesterol places individuals and populations at lower risk. Because of the high cost, insurance concerns and suboptimal access to physician care, a self-directed, effective and safe approach to cholesterol maintenance or reduction would be very desirable. Drug therapy also has been associated with suboptimal results. Though a new concept that addresses cholesterol by several mechanisms simultaneously has been shown to be more consistently effective and with better tolerability, there is still a need for a self-directed cholesterol optimizing alternative. It is, therefore, our intent in this study to evaluate certain foods, specifically nutraceutical containing fruit flavored drinks in the hopes that they can be proven a safe and effective alternative approach for cholesterol management.

DETAILED DESCRIPTION:
Cholesterol is the principle component of cardiovascular disease. It deposits in the walls of blood vessels and contributes to both chronic vascular insufficiency manifested as claudication, ischemic ulceration, or angina, and acute vascular insufficiency presenting as heart attack, stroke or sudden death.

Coronary heart disease is the number one killer worldwide. Approximately 50% of males and one-third of females will develop a coronary heart disease related acute event in their lifetime. The cost of coronary heart disease is staggering. In the United States alone, over $120 billion is spent annually in direct and indirect costs attributed to this killer (10).

The Framingham Heart Study has shown that coronary heart disease incidence rises proportionately to serum cholesterol (1). More importantly, numerous studies demonstrate a reduction in coronary heart disease related events with falling cholesterol levels on treatment (18).

There are four classes of commonly used cholesterol lowering drugs:

1. statins
2. fibric acid derivates
3. niacin
4. bile acid sequestrants.

Of these, the most widely used are the statins. Statins produce potent LDL lowering, reduce cardiovascular events, and are relatively safe. However, despite their proven effectiveness and relative safety, even statins have their limitations. First, as many as 30% of people who take statins develop myalgias. Second, many drug interactions exist. Third, most of the LDL lowering is seen with the lowest dose, making up-titration of limited value (3) (20). With fibrates, niacin, and bile acid sequestrants, tolerability is even more problematic with titration, and end point data somewhat weaker than with statins, especially for monotherapy (4)(7)(14)(17).

Beyond the efficacy and safety limitations of the selected drug, there are socioeconomic barriers to effective cholesterol lowering. Although people are cognizant of the importance of cholesterol reduction, many evade the doctor/patient relationship at all cost. Others do not like, forget to take, or have difficulty swallowing pills. Some do not have access to health care, drug plans, or lack the financial means to afford pharmaceuticals. Furthermore, high cholesterol represents a label that might adversely affect one's ability to procure inexpensive life and health insurance. Therefore, there is a need for alternative cholesterol lowering approaches that circumvent these limitations.

In devising these approaches, it is crucial to incorporate a relatively new concept in cholesterol lowering and/or maintenance. Recently, it has become apparent that targeting a single mechanism, either of absorption or endogenous production of cholesterol, may augment the other potentially compensatory mechanism, thus decreasing the effectiveness of any type of monotherapy. Hence, raising the dose of any one medication may enhance toxicity out of proportion to any gain in efficacy. To be effective without substantial toxicity, several medications or active ingredients that lower cholesterol via different mechanisms should be employed simultaneously. The rationale for this application has been tested and proven for combination statin/niacin therapy (12) (15) (22) and also combination statin/phytosterol therapy (16). In each case, the reduction from combination therapy is greater than that expected from the sum reductions of the constituents, thereby, allowing for lower doses of drugs and lower toxicity compared to single drug therapy (21).

There are several non-pharmaceutical products available to the public that have cholesterol lowering properties; L-carnitine and vitamin C are two such examples, and these substances are thought completely safe at the low dose ranges shown effective for cholesterol lowering. L-carnitine facilitates fatty acid transfer and intracellular mitochondrial metabolism, removing cholesterol from the blood and thereby reducing serum cholesterol. Though side effects are very rare and dose related, lowering of seizure threshold in patients with a history of seizures has been reported (5) (8). Vitamin C has statin-like HMG-coA reductase inhibitory activity, but unlike statins, lowers cholesterol without raising LPa or depleting Co-enzyme Q-10 (two counterproductive effects of statins). Vitamin C has been shown completely safe to a dosage of 3 grams per day (9).

Co-Q-10 has been demonstrated to mitigate the side effects of statins (myalgias) and its depletion may reduce cardiac muscle function. Side effects of Co-Q-10 are rare and usually involve skin irritation so minor GI side effects (19).

Red Yeast Rice is a Chinese dietary supplement available as a flavoring and coloring agent for centuries. It is known to contain at least nine different statins as well as phytosterols. Thus, it decreases both the body's synthesis of cholesterol and its absorption. Though the form augmented for Lovastatin content is illegal in the United States, the naturally fermented product is available legally at health food stores to promote favorable cholesterol levels. The red coloration may also stimulate appetite and hence compliance with food or dietary supplements that contain it. Though Red Yeast Rice is, in general, well-tolerated, headache, GI side effects, muscle pain or weakness, liver abnormalities and dizziness have rarely been reported. The psychological benefit of enhanced compliance through the red coloration of Red Yeast Rice may be further augmented by L-carnitine, which has been shown to stimulate a mild sense of euphoria (2) (11).

Niacin is a B vitamin that lowers LDL and triglycerides and raises HDL, in part, by decreasing the hepatic release of lipoproteins that bind cholesterol. Though comparatively high doses of niacin are often needed to lower LDL, the beneficial effects on HDL have been realized on very low doses. Though greater than 2 grams, predominantly of the long-acting niacin formulation, have been associated with side effects including flushing, GI side effects, hyperglycemia, gout, abnormal liver function and myopathy. Very low doses of niacin are very well-tolerated (22).

Phytosterols are natural plant products that lower cholesterol by competing with cholesterol for absorption in the intestine (13). The data in support for cholesterol reduction and cardiovascular health improvement is so strong that the FDA allows products that contain sufficient quantities of phytosterols to make special claims concerning cardiovascular benefits (6). Very well-tolerated, up to 3 grams per day, is thought to be essentially devoid of side effects (13).

An ideal cholesterol lowering product would be proven effective, and with minimal side effects. It would not require one to take pills, and would preferably be in liquid form as a suspension or soluble drink. It would contain multiple active ingredients that would work by different mechanisms at different sites to allow a lower side effect profile with synergistic efficacy.

ELIGIBILITY:
Inclusion Criteria:

All subjects will need to be on their usual diet and

1. Not have been on any cholesterol lowering medications for at least two months or eight weeks prior to randomization. The subjects will also need to be off of all dietary supplements or vitamins containing any of the constituents in any of the formulations for the same time period.
2. Any baseline cholesterol measurement will be acceptable since there is no convincing evidence of low cholesterol below which a clinical benefit is thought not to occur, nor cellular function compromised,.
3. Males 20 to 80 years of age will be acceptable.
4. Post menopausal females 55 to 80 years of age.

Exclusion Criteria:

1. Prior myocardial infarction clinically or by EKG criteria including left bundle branch block.
2. History of angina.
3. History of abnormal stress test consistent with ischemia or myocardial infarction.
4. Diabetes (because of the generally accepted significant association with previously undiagnosed coronary artery disease).
5. Peripheral vascular disease (because of the generally accepted significant association with previously undiagnosed coronary artery disease).
6. History of prior allergy or sensitivity to any component of any formulation.
7. Those taking medications of the following types or closely related medications:

   1. cyclosporins
   2. fibrates
   3. Azole antifungals
   4. macrolide antibiotics
   5. anti-arrhythmic medications
   6. Nefazodin
   7. protease inhibitors
   8. Coumadin
   9. Seizure medication
8. Pre-randomization CPK greater than the upper limits of normal.
9. History of hepatitis or unexplained elevation of transaminase LFTs.
10. History of musculoskeletal condition with weakness or pain, i.e., arthritis, myositis, myalgia, fibromyalgia or PMR.
11. Active cancer or vasculitis on therapy.
12. Inability to provide informed consent.
13. Premenopausal women, women who are pregnant, may become pregnant or nursing mothers will be excluded because of the unknown effects of nutraceuticals on the fetus or newborn.
14. Any travel plans by the subject that would affect compliance with the study protocol.
15. History of a seizure disorder.
16. End stage renal disease (or renal failure).
17. Any subject who the investigator determines that discontinuing current cholesterol lowering treatment for the 16 weeks (8 weeks each for a wash out and study participation) of the study would not be safe or otherwise in the best interest of the subject.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
LDL Reduction | 8 weeks
  The primary end point will be relative LDL and total cholesterol reductions, i.e., the placebo subtracted reduction in these parameters.

SECONDARY OUTCOMES:
HDL change from control formulation | 8 weeks
  Secondary end points will include change from the control formulation with regard to HDL.
CRP change from control formulation | 8 weeks
  Secondary end points will include change from the control formulation with regard to CRP.
Triglyceride reduction from control formulation | 8 weeks
  Secondary end points will include change from the control formulation with regard to triglyceride levels.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Karl, M.D., Principal Investigator — Boca Raton Community Hospital
Locations (1):
- Mitchell Karl, M.D. -- Cardiology, Boca Raton, Florida, United States

REFERENCES:
- [Background] Abbott R.D., McGee, D., The Framingham Study, Section 37. The Probability Of Developing Certain Cardiovascular Diseases In Eight Years At Specified Values Of Some Characteristics. NIH publication #No. 87-2284. Washington: Government Printing Office, 1987.
- [Background] Baens-Arcega, L., Ardischer, AG et al. Indigenous Amino Acid/Peptide Sauces and Pastes with Meat-Like Flavors, Chinese Soy Sauces, Japanese, Shoyu, Japanese Miso, Southeast Asian Fish Sauces and Pastes and Related Fermented Foods in: Steinkraus, ED Handbook of Indigenous Fermented Food, 2nd edition, New York, NY, Marcel Dekker, Inc., 1986. Pg 625-633.
- [Background] Bellosta S, Paoletti R, Corsini A. Safety of statins: focus on clinical pharmacokinetics and drug interactions. Circulation. 2004 Jun 15;109(23 Suppl 1):III50-7. doi: 10.1161/01.CIR.0000131519.15067.1f. PMID 15198967
- [Background] Brown G, Albers JJ, Fisher LD, Schaefer SM, Lin JT, Kaplan C, Zhao XQ, Bisson BD, Fitzpatrick VF, Dodge HT. Regression of coronary artery disease as a result of intensive lipid-lowering therapy in men with high levels of apolipoprotein B. N Engl J Med. 1990 Nov 8;323(19):1289-98. doi: 10.1056/NEJM199011083231901. PMID 2215615
- [Background] Diaz, et al, L-Carnitine Induced Modulation of Plasma Fatty Acid Metabolism, Rev Electron J. BioMed 2006; 1:33.
- [Background] FDA Authorizes New Coronary Heart Disease Health Claims for Plant Sterols and Plant Stanol Esters". FDA Talk Paper, 09/05/2000, Available at http://www.cfsan.fda.gov/ird/ttsterol.html.
- [Background] Frick MH, Elo O, Haapa K, Heinonen OP, Heinsalmi P, Helo P, Huttunen JK, Kaitaniemi P, Koskinen P, Manninen V, et al. Helsinki Heart Study: primary-prevention trial with gemfibrozil in middle-aged men with dyslipidemia. Safety of treatment, changes in risk factors, and incidence of coronary heart disease. N Engl J Med. 1987 Nov 12;317(20):1237-45. doi: 10.1056/NEJM198711123172001. PMID 3313041
- [Background] FRITZ IB. CARNITINE AND ITS ROLE IN FATTY ACID METABOLISM. Adv Lipid Res. 1963;1:285-334. No abstract available. PMID 14248955
- [Background] Harwood HJ Jr, Greene YJ, Stacpoole PW. Inhibition of human leukocyte 3-hydroxy-3-methylglutaryl coenzyme A reductase activity by ascorbic acid. An effect mediated by the free radical monodehydroascorbate. J Biol Chem. 1986 Jun 5;261(16):7127-35. PMID 3711081
- [Background] Rosamond W, Flegal K, Friday G, Furie K, Go A, Greenlund K, Haase N, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell CJ, Roger V, Rumsfeld J, Sorlie P, Steinberger J, Thom T, Wasserthiel-Smoller S, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2007 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2007 Feb 6;115(5):e69-171. doi: 10.1161/CIRCULATIONAHA.106.179918. Epub 2006 Dec 28. No abstract available. PMID 17194875
- [Background] Heber D, Yip I, Ashley JM, Elashoff DA, Elashoff RM, Go VL. Cholesterol-lowering effects of a proprietary Chinese red-yeast-rice dietary supplement. Am J Clin Nutr. 1999 Feb;69(2):231-6. doi: 10.1093/ajcn/69.2.231. PMID 9989685
- [Background] Insull W Jr, McGovern ME, Schrott H, Thompson P, Crouse JR, Zieve F, Corbelli J. Efficacy of extended-release niacin with lovastatin for hypercholesterolemia: assessing all reasonable doses with innovative surface graph analysis. Arch Intern Med. 2004 May 24;164(10):1121-7. doi: 10.1001/archinte.164.10.1121. PMID 15159270
- [Background] Katan MB, Grundy SM, Jones P, Law M, Miettinen T, Paoletti R; Stresa Workshop Participants. Efficacy and safety of plant stanols and sterols in the management of blood cholesterol levels. Mayo Clin Proc. 2003 Aug;78(8):965-78. doi: 10.4065/78.8.965. PMID 12911045
- [Background] Keech A, Simes RJ, Barter P, Best J, Scott R, Taskinen MR, Forder P, Pillai A, Davis T, Glasziou P, Drury P, Kesaniemi YA, Sullivan D, Hunt D, Colman P, d'Emden M, Whiting M, Ehnholm C, Laakso M; FIELD study investigators. Effects of long-term fenofibrate therapy on cardiovascular events in 9795 people with type 2 diabetes mellitus (the FIELD study): randomised controlled trial. Lancet. 2005 Nov 26;366(9500):1849-61. doi: 10.1016/S0140-6736(05)67667-2. PMID 16310551
- [Background] McKenney JM, Jones PH, Bays HE, Knopp RH, Kashyap ML, Ruoff GE, McGovern ME. Comparative effects on lipid levels of combination therapy with a statin and extended-release niacin or ezetimibe versus a statin alone (the COMPELL study). Atherosclerosis. 2007 Jun;192(2):432-7. doi: 10.1016/j.atherosclerosis.2006.11.037. Epub 2007 Jan 19. PMID 17239888
- [Background] Radermecker RP, Scheen AJ. Serum plant sterols and atherosclerosis: is there a place for statin-ezetimibe combination? J Am Coll Cardiol. 2006 Apr 4;47(7):1496-7; author reply 1497-8. doi: 10.1016/j.jacc.2006.01.031. Epub 2006 Mar 20. No abstract available. PMID 16580546
- [Background] Morris DL, Kritchevsky SB, Davis CE. Serum carotenoids and coronary heart disease. The Lipid Research Clinics Coronary Primary Prevention Trial and Follow-up Study. JAMA. 1994 Nov 9;272(18):1439-41. doi: 10.1001/jama.272.18.1439. PMID 7933426
- [Background] Muldoon MF, Manuck SB, Matthews KA. Lowering cholesterol concentrations and mortality: a quantitative review of primary prevention trials. BMJ. 1990 Aug 11;301(6747):309-14. doi: 10.1136/bmj.301.6747.309. PMID 2144195
- [Background] Mortensen SA. Perspectives on therapy of cardiovascular diseases with coenzyme Q10 (ubiquinone). Clin Investig. 1993;71(8 Suppl):S116-23. doi: 10.1007/BF00226851. PMID 8241694
- [Background] Pasternak RC, Smith SC Jr, Bairey-Merz CN, Grundy SM, Cleeman JI, Lenfant C; American College of Cardiology; American Heart Association; National Heart, Lung and Blood Institute. ACC/AHA/NHLBI Clinical Advisory on the Use and Safety of Statins. Circulation. 2002 Aug 20;106(8):1024-8. doi: 10.1161/01.cir.0000032466.44170.44. No abstract available. PMID 12186811
- [Background] Schectman G, Hiatt J. Dose-response characteristics of cholesterol-lowering drug therapies: implications for treatment. Ann Intern Med. 1996 Dec 15;125(12):990-1000. doi: 10.7326/0003-4819-125-12-199612150-00011. PMID 8967711
- [Background] Wink J, Giacoppe G, King J. Effect of very-low-dose niacin on high-density lipoprotein in patients undergoing long-term statin therapy. Am Heart J. 2002 Mar;143(3):514-8. doi: 10.1067/mhj.2002.120158. PMID 11868059
- [Background] Shin MJ, Lee JH, Jang Y, Lee-Kim YC, Park E, Kim KM, Chung BC, Chung N. Micellar phytosterols effectively reduce cholesterol absorption at low doses. Ann Nutr Metab. 2005 Sep-Oct;49(5):346-51. doi: 10.1159/000087880. Epub 2005 Aug 26. PMID 16127299
- [Background] The Lipid Research Clinics Coronary Primary Prevention Trial results. II. The relationship of reduction in incidence of coronary heart disease to cholesterol lowering. JAMA. 1984 Jan 20;251(3):365-74. PMID 6361300
- [Background] Thompson GR, O'Neill F, Seed M. Why some patients respond poorly to statins and how this might be remedied. Eur Heart J. 2002 Feb;23(3):200-6. doi: 10.1053/euhj.2001.3071. No abstract available. PMID 11792134